CLINICAL TRIAL: NCT02376556
Title: The Prevalence of Dry Eye Syndrome Among Patients Who Underwent Upper Eyelids Blepharoplasty With and Without Muller Muscle Resection
Brief Title: The Effect of Eyelid Surgery on Dry Eye - a Prospective Study
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Guy Ben Simon, Head, Orbital, Ophthalmic Plastic & Lacrimal Surgery department, The Goldschleger Eye Institute, Sheba Medical Center, Tel Hashomer, Israel, Sheba Medical Center
Other Study IDs: SHEBA-14-1496-GBS-CTIL
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye Syndrome; Ptosis; Dermatochalasis
Keywords: Dry eye syndrome; Blepharoplasty; Muller muscle resection surgery
MeSH Terms: conditions — Dry Eye Syndromes; Blepharoptosis; Cutis Laxa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blepharoplasty: patients undergoing upper eyelid blepharoplasty
- blepharoplasty and muller muscle resection: patients undergoing a combined blepharoplasty and muller muscle resection surgery

SUMMARY:
The investigators aim to assess the effect of blepharoplasty with or without muller muscle resection on the symptoms of dry eye syndrome. this will be an observational study in which patients undergoing the aforementioned surgeries will be followed up and monitored for dry eye symptoms.

DETAILED DESCRIPTION:
Patients who are referred for blepharoplasty with or without muller muscle resection in the oculoplastic clinic in the investigators institution, will be offered to participate in the study. After filling and informed consent form, patients recruited will fill in a questionnaire about dry eye symptoms, and will be examined by an ophthalmologist for visual acuity, intra ocular pressure, anterior segment examination using a slit lamp biomicroscopy, schirmer test, tear break up time assessment and tear osmolarity. These are all standard examination in ophthalmology. The surgical procedure planned to correct the eyelid pathology will not be affected by the results of these examinations.

The same combination of ophthalmic examination will by done on postoperative follow-up examination 1 week, 1 month and 3 months after the surgery. Dry eye questionnaire will be filled in by the patients on postoperative follow-up examination 1 month and 3 months after the surgery.

This data will help us assess the effect of these common surgical procedures on dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

* patients who are referred for blepharoplasty with or without muller muscle resection in the oculoplastic clinic in our institution
* no other ophthalmic procedures planned for the patient in study period
* ability to undergo full ophthalmic examination as stated in the study protocol
* Ability to complete the dry eye questionnaire
* ability to sign an informed consent form

Exclusion Criteria:

* previous eyelid surgery
* other orbital or lacrimal gland disease
* concurrent use of contact lenses
* concurrent use of Restasis
* previous glaucoma surgery
* use of punctual plugs
* pregnant or nursing women

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are referred for blepharoplasty with or without muller muscle resection in the oculoplastic clinic in our institution
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Objective assessment of dry eye syndrome | 3 months postoperatively

SECONDARY OUTCOMES:
Subjective assessment of dry eye syndrome | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Guy J Ben Simon, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel